CLINICAL TRIAL: NCT05369494
Title: Tolerance of Infants Fed a Hydrolyzed Infant Formula
Brief Title: Infants Fed a Hydrolyzed Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AL49
Record Dates: First submitted 2022-05-03; First posted 2022-05-11 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Gastrointestinal Tolerance
MeSH Terms: interventions — Oligosaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Product (Experimental): Infant formula product consumed ad libitum as instructed for approximately 28 days; Powder formula mixed to 20 kcal/fl. oz.
  Interventions: Other: Hydrolyzed protein infant formula with oligosaccharides

INTERVENTIONS:
Other: Hydrolyzed protein infant formula with oligosaccharides — Hydrolyzed protein infant formula with oligosaccharides

SUMMARY:
The purpose of this non-randomized, multi-center study is to evaluate the growth, tolerance and compliance of an extensively hydrolyzed infant formula in an intended use population of infants.

ELIGIBILITY:
Inclusion Criteria:

* Infant is 0 to 90 days of age at enrollment.
* Formula-fed Infant who is either experiencing persistent feeding intolerance, symptoms of suspected food protein allergy or currently consuming an extensively hydrolyzed formula (EHF) for symptoms of suspected food protein allergy, persistent feeding intolerance symptoms or other conditions where EHF is deemed an appropriate feeding by their health care professional
* Parent(s) of infants confirm their intention not to administer prescription medications, OTC medications, home remedies, prebiotics, probiotics, herbal preparations or rehydration fluids that might affect GI tolerance, unless their infants are currently consuming and have been directed by their healthcare professional to continue their use during the study
* Parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study.
* Parent(s) confirm their intention not to administer solid foods or juices to their infant from enrollment through the duration of the study
* Parent(s) confirm their intention not to administer vitamin or mineral supplements (with the exception of Vitamin D supplements) to their infant from enrollment through the duration of the study, unless instructed otherwise by their healthcare professional
* Infant's parent(s) or a LAR has voluntarily signed and dated an informed consent form (ICF) approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study

Exclusion Criteria:

* An adverse maternal, fetal or participant medical history that is thought by the investigator to have potential for effects on growth, and/or development
* Awareness of a positive drug screen in the mother or participant
* Suspected maternal substance abuse including alcohol
* Participation in another study that has not been approved as a concomitant study by AN
* Participant is receiving oral or inhaled steroids
* Participant has an allergy or intolerance to any ingredient in the study product, as reported by the parent
* Participant has received an amino acid-based formula

Ages: 0 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
Weight Maintenance | Study Day1 to Study Day 28
  Change in weight for age z-score

SECONDARY OUTCOMES:
Gastrointestinal Tolerance | Study Day1 to Study Day 28
  Parent completed diary
Weight | Study Day1 to Study Day 28
  Weight gain per day in grams
Length | Study Day1 to Study Day 28
  Length gain per day in cm

OTHER OUTCOMES:
Parent Perspectives Questionnaire | Study Day1 to Study Day 28
  Parent completed questionnaire; 4, 5-point Likert scale questions, scaled from negative to positive with higher scores indicating better perception
Formula Satisfaction Questionnaire | Study Day1 to Study Day 28
  Parent completed questionnaire; 13 questions of up to 5 categories, scaled from positive to negative
Infant Feeding and Stool Patterns Questionnaire | Study Day1 to Study Day 28
  Parent completed questionnaire; 16, 5-point Likert scale questions, scaled from always to never
Health Care Utilization | Study Day1 to Study Day 28
  Number of Visits
Adverse Events | Study Day1 to Study Day 28
  Parent reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Carlett Ramirez, Study Chair — Abbott Nutrition
Locations (7):
- United States (7):
  - Meridian Clinical Research, LLC, Washington D.C., District of Columbia
  - AdventHealth Medical Group Pediatrics, Orange City, Florida
  - Javara Inc., Fayetteville, Georgia
  - Meridian Clinical Research 3259, Macon, Georgia
  - Springs Medical Research, Owensboro, Kentucky
  - Meridian Clinical Research 3357, Charleston, South Carolina
  - Gentle Pediatrics, Houston, Texas

IPD SHARING:
Plan to Share IPD: No